CLINICAL TRIAL: NCT04723394
Title: A Phase III Randomized, Double-blind, Placebo-controlled, Multicenter Study to Determine the Safety and Efficacy of AZD7442 for the Treatment of COVID-19 in Non-hospitalized Adults
Brief Title: Phase III Study of AZD7442 for Treatment of COVID-19 in Outpatient Adults
Acronym: TACKLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D8851C00001
Record Dates: First submitted 2021-01-14; First posted 2021-01-25 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
Keywords: Treatment of COVID-19
MeSH Terms: conditions — COVID-19 | interventions — cilgavimab and tixagevimab drug combination; tixagevimab; cilgavimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD7442 (Experimental): Up to approximately 1700 participants will be randomized in a 1:1 ratio. Arm 1 (n=up to approximately 850) will receive a single dose (× 2 IM injections) of 600 mg of AZD7442.
  Interventions: Drug: AZD7442
- Placebo (Placebo Comparator): Up to approximately 1700 participants will be randomized in a 1:1 ratio. Arm 2 (n=up to approximately 850) will receive saline placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7442 — Single dose (× 2 separate IM injections) of 600 mg of AZD7442 or saline placebo on Day 1.
  Other Names: Combination of 2 mAbs (AZD8895 and AZD1061)
  Arms: AZD7442
Drug: Placebo — Single dose (× 2 separate IM injections) of 600 mg of AZD7442 or saline placebo on Day 1.
  Arms: Placebo

SUMMARY:
This Phase III study will assess whether AZD7442 (a combination of 2 mAbs) can safely treat outpatient adults with COVID-19 and prevent either severe COVID-19 or death.

DETAILED DESCRIPTION:
A novel coronavirus, SARS-CoV-2, first emerged in China in November 2019 causing cases of atypical pneumonia. As of 6 October 2020, the virus has spread to all corners of the globe, with over 35 million confirmed cases reported and more than one million associated deaths according to the WHO. The COVID-19 pandemic is causing major disruption to global healthcare systems with significant socioeconomic impacts. Effective interventions to prevent or treat COVID-19 remain few in number and clinical experience is limited.

There is an urgent need to rapidly evaluate treatments in the non-hospitalized setting to prevent progression and reduce serious complications of COVID-19, as well as its transmission.

As a response to the ongoing pandemic, AstraZeneca is developing mAbs to the SARS-CoV-2 spike protein. The SARS-CoV-2 spike protein contains the virus's RBD, which enables the virus to bind to receptors on human cells. By targeting this region of the virus's spike protein, antibodies can block the virus's attachment to human cells, and, therefore, is expected to block infection. Amino acid substitutions have been introduced into the antibodies to both extend their half-lives, which should prolong their potential prophylactic benefit, and decrease Fc effector function in order to decrease the potential risk of antibody-dependent enhancement of disease.

AZD7442, a combination of 2 of these mAbs (AZD8895 and AZD1061), is being evaluated for administration to treat or prevent COVID-19. There are currently one ongoing Phase I study and two ongoing Phase III studies with AZD7442, in addition to this treatment study.

Enrollment of up to approximately 1700 participants is planned.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has a documented laboratory-confirmed SARS-CoV-2 infection, as determined by a molecular test (antigen or nucleic acid) from any respiratory tract specimen (eg, oropharyngeal, NP, or nasal swab, or saliva) collected ≤ 3 days prior to Day 1.
2. WHO Clinical Progression Scale score > 1 and < 4.
3. Participant must be dosed with IMP no more than 7 days from self-reported onset of COVID-19-related symptoms (mild to moderate COVID-19) or measured fever, defined as the self-reported date of first reported sign/symptom.
4. One or more of the following signs/symptoms must be present within 24 hours prior to Day1: Cough, Sore throat, Shortness of breath or difficulty breathing at rest or with activity, Body pain or muscle pain/aches, Fatigue, Headache, Chills, Nasal obstruction or congestion, Nasal discharge, Nausea or vomiting, Diarrhea, New loss of taste or smell.
5. Oxygenation saturation of ≥ 92% obtained at rest by study staff within 24 hours prior to Day 1 (unless participant regularly receives chronic supplementary oxygen for an underlying lung condition).
6. Participant agrees not to participate in another clinical trial for the treatment of COVID-19 or SARS-CoV-2 during the study period until reaching hospitalization or 28 days after entry into the study (whichever is earliest).
7. Participant must be ≥ 18 years of age, provide informed consent and is able to comply with study requirements/procedures.
8. Male participants: Contraception for male participants is not required; however, to avoid the transfer of any fluids, all male participants must use a condom from Day 1 and agree to continue through 90 days following administration of IMP.
9. Women of childbearing potential must use one highly effective form of birth control.

Exclusion Criteria:

1. History or current hospitalization for COVID-19.
2. Current need for hospitalization/immediate medical attention in a clinic/emergency room service
3. Previous hypersensitivity, infusion related reaction, or adverse reaction to any monoclonal antibodies or known allergy to components of the IMP or placebo.
4. Receipt of any investigational or licensed vaccine for prevention of COVID-19 at any time prior to entry into this study or expected administration immediately after enrollment.
5. Current requirement or anticipated impending need for mechanical ventilation.
6. Any significant disease, disorder or finding that may increase risk to the participant that might affect his/her ability to participate in this study.
7. Received convalescent COVID-19 plasma treatment any time prior to entry into this study.
8. Receipt of systemic steroids (e.g., prednisone, dexamethasone) or inhaled steroids within 30 days prior to study entry, unless a stable dose is used for a chronic condition.
9. Receipt of any IMP in the previous 90 days or 5 half lives (whichever is longer), or expected receipt of IMP during the study follow-up period, or concurrent participation in another interventional study.
10. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 910 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-08-21 (Actual); Study Completion 2022-10-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (89):
- United States (20):
  - Research Site, Jasper, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Long Beach, California
  - Research Site, Northridge, California
  - Research Site, Cutler Bay, Florida
  - Research Site, Miami, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Lake Charles, Louisiana
  - Research Site, St Louis, Missouri
  - Research Site, La Vista, Nebraska
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Columbus, Ohio
  - Research Site, West Columbia, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Humble, Texas
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Munro
- Brazil (5):
  - Research Site, Blumenau
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São Paulo
  - Research Site, Sorocaba
- Czechia (3):
  - Research Site, Hradec Králové
  - Research Site, Kolín
  - Research Site, Svitavy
- Germany (11):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Friedrichshain
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Koblenz
  - Research Site, Mainz
  - Research Site, München
  - Research Site, München-Pasing
- Hungary (2):
  - Research Site, Debrecen
  - Research Site, Gyöngyös
- Italy (5):
  - Research Site, Guastalla
  - Research Site, Milan
  - Research Site, Piacenza
  - Research Site, Pisa
  - Research Site, Roma
- Japan (9):
  - Research Site, Chiba
  - Research Site, Hachioji-shi
  - Research Site, Iruma-Gun
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Narita-shi
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
- Mexico (9):
  - Research Site, Chihuahua City
  - Research Site, Cuauhtémoc
  - Research Site, Cuautitlán Izcalli
  - Research Site, Ecatepec de Morelos
  - Research Site, Guadalajara
  - Research Site, Mazatlán
  - Research Site, Mérida
  - Research Site, Monterrey
  - Research Site, Tlalpan
- Research Site, Lima, Peru
- Poland (2):
  - Research Site, Rzeszów
  - Research Site, Wołomin
- Russia (3):
  - Research Site, Moscow
  - Research Site, Murmansk
  - Research Site, Saint Petersburg
- Spain (5):
  - Research Site, Cabra
  - Research Site, Centelles (Barcelona)
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Málaga
- Ukraine (3):
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kherson
- United Kingdom (9):
  - Research Site, Blackpool
  - Research Site, Bracknell
  - Research Site, Bristol
  - Research Site, Cambridge
  - Research Site, Connor Downs
  - Research Site, Highgate
  - Research Site, Leicester
  - Research Site, Preston
  - Research Site, Rochdale

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Ashraf-Kashani and Kumar 2017 Ashraf-Kashani N, Kumar R. High-flow nasal oxygen therapy. BJA Education. 2017;17:57-62.
- [Background] Gou and Xi 2019 Gou J, Xi D. Hierarchical testing of a primary and a secondary endpoint in a group sequential design with different information times. Statistics in Biopharmaceutical Research. 2019;11(4):398-406, DOI: 10.1080/19466315.2018.1546613.
- [Background] ICMRA 2020 International Coalition of Medicines Regulatory Authorities. Global regulatory workshop on COVID-19 therapeutics: agreement on acceptable endpoints for clinical trials. Published online July 2020. Retrieved from http://icmra.info/drupal/news/20july2020/summary
- [Background] Li F. Structure, Function, and Evolution of Coronavirus Spike Proteins. Annu Rev Virol. 2016 Sep 29;3(1):237-261. doi: 10.1146/annurev-virology-110615-042301. Epub 2016 Aug 25. PMID 27578435
- [Background] Miettinen O, Nurminen M. Comparative analysis of two rates. Stat Med. 1985 Apr-Jun;4(2):213-26. doi: 10.1002/sim.4780040211. PMID 4023479
- [Background] Sharma S, Danckers M, Sanghavi DK, Chakraborty RK. High-Flow Nasal Cannula. 2023 Apr 6. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK526071/ PMID 30252327
- [Background] Tamhane AC, Mehta CR, Liu L. Testing a primary and a secondary endpoint in a group sequential design. Biometrics. 2010 Dec;66(4):1174-84. doi: 10.1111/j.1541-0420.2010.01402.x. PMID 20337631
- [Background] WHO 2020 WHO COVID-19 Dashboard. Available from: https://covid19.who.int
- [Background] WHO Working Group on the Clinical Characterisation and Management of COVID-19 infection. A minimal common outcome measure set for COVID-19 clinical research. Lancet Infect Dis. 2020 Aug;20(8):e192-e197. doi: 10.1016/S1473-3099(20)30483-7. Epub 2020 Jun 12. PMID 32539990
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Zou G. A modified poisson regression approach to prospective studies with binary data. Am J Epidemiol. 2004 Apr 1;159(7):702-6. doi: 10.1093/aje/kwh090. PMID 15033648
- [Background] CDC, 2021 CDC, Investigating the Impact of COVID-19 during Pregnancy, available from https://www.cdc.gov/coronavirus/2019-ncov/cases-updates/special-populations/pregnancy-data-on-covid-19/what-cdc-is-doing.html
- [Background] CDC, Growth Charts CDC, Growth Charts, available from https://www.cdc.gov/growthcharts/clinical_charts.htm
- [Background] Lilly BLAZE-1 2021 Lilly. Lilly's bamlanivimab and etesevimab together reduced hospitalizations and death in Phase 3 trial for early COVID-19. Published online 10 March 2021. Accessed 31 March 2021. https://investor.lilly.com/news-releases/news-release-details/lillys-bamlanivimab-and-etesevimab-together-reduced
- [Background] Regeneron Pharmaceuticals, Inc. REGEN-COV Outpatient Trial 2021 Regeneron Pharmaceuticals, Inc. Phase 3 trial shows Regen-Cov™ (casirivimab with imdevimab) antibody cocktail reduced hospitalization or death by 70% in non-hospitalized Covid-19 patients. Published online 23 March 2021. Accessed 31 March 2021. https://investor.regeneron.com/news-releases/news-release-details/phase-3-trial-shows-regen-covtm-casirivimab-imdevimab-antibody#:~:text=This%20definitive%20Phase%203%20outcomes,71%25%20(2%2C400%20mg%20IV)
- [Derived] Hobbs FDR, Montgomery H, Padilla F, Simon-Campos JA, Arbetter D, Seegobin S, Kiazand A, Streicher K, Martinez-Alier N, Cohen TS, Esser MT. Safety, Efficacy and Pharmacokinetics of AZD7442 (Tixagevimab/Cilgavimab) for Treatment of Mild-to-Moderate COVID-19: 15-Month Final Analysis of the TACKLE Trial. Infect Dis Ther. 2024 Mar;13(3):521-533. doi: 10.1007/s40121-024-00931-4. Epub 2024 Feb 25. PMID 38403865
- [Derived] Hobbs FDR, Montgomery H, Padilla F, Simon-Campos JA, Kim K, Arbetter D, Padilla KW, Reddy VP, Seegobin S, Streicher K, Templeton A, Viani RM, Johnsson E, Koh GCKW, Esser MT. Outpatient Treatment with AZD7442 (Tixagevimab/Cilgavimab) Prevented COVID-19 Hospitalizations over 6 Months and Reduced Symptom Progression in the TACKLE Randomized Trial. Infect Dis Ther. 2023 Sep;12(9):2269-2287. doi: 10.1007/s40121-023-00861-7. Epub 2023 Sep 26. PMID 37751015
- [Derived] Montgomery H, Hobbs FDR, Padilla F, Arbetter D, Templeton A, Seegobin S, Kim K, Campos JAS, Arends RH, Brodek BH, Brooks D, Garbes P, Jimenez J, Koh GCKW, Padilla KW, Streicher K, Viani RM, Alagappan V, Pangalos MN, Esser MT; TACKLE study group. Efficacy and safety of intramuscular administration of tixagevimab-cilgavimab for early outpatient treatment of COVID-19 (TACKLE): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Respir Med. 2022 Oct;10(10):985-996. doi: 10.1016/S2213-2600(22)00180-1. Epub 2022 Jun 7. PMID 35688164
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8851C00001&attachmentIdentifier=dd6cb212-7d2d-40c2-a4b9-39d661461486&fileName=Clinical_Study_Protocol_Redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8851C00001&attachmentIdentifier=7e4b7190-a3a8-49b7-8cce-8d5b0c3da7ae&fileName=Statistical_Analysis_Plan__Redacted.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8851C00001&attachmentIdentifier=a1495ac4-8d00-4c45-b026-1f0084417cb8&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 910 participants were randomized to receive treatment in study D8851C00001 (TACKLE) with AZD7442 (AZD8895 + AZD1061) or placebo. Of the 910 participants randomized, 903 (99.2%) received treatment with study drug. Of the 903 dosed, 452 (50.1%) participants received AZD7442 and 451 (49.9%) participants received placebo.
Pre-assignment Details: In TACKLE, at the first visit, ie, the enrollment visit 1, participants were evaluated regarding the protocol mandated inclusion and exclusion criteria. After enrolment, eligible participants were randomized at a 1: 1 ratio to receive a single dose of study provided AZD7442 (AZD8895 + AZD1061) or placebo.
Groups:
- AZD7442: Single dose of 600 mg of AZD7442 (2 separate IM injections) on Day 1
- Placebo: Single dose of Placebo (2 separate IM injections) on Day 1
Period: Overall Study
Arm/Group | AZD7442 | Placebo
Started (All Participants Randomized) | 456 | 454
Dosed (Full Analysis Set) | 452 | 451
Modified Full Analysis Set (Dosed, randomized <=7 days from symptom onset and not hospitalized for isolation purposes at baseline) | 413 | 421
Primary Analysis Population (Participants who are included in the modified full analysis set excluding those who did not have an assessment for the primary endpoint) | 410 | 419
Key Secondary Analysis Population (Participants who are included in the modified full analysis set excluding those who did not have an assessment for the key secondary endpoint) | 404 | 411
Completed | 407 | 390
Not Completed | 49 | 64
Not completed — Adverse Event | 0 | 3
Not completed — Death | 8 | 8
Not completed — Lost to Follow-up | 20 | 17
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 20 | 34
Not completed — Participants withdrawn due to eligibility, eligibility, moving, and being randomized in error. | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set - All participants randomized and dosed with IMP
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD7442 | Placebo | Total
Number analyzed (Participants) | 452 | 451 | 903
Age, Continuous [Median (Full Range); unit: Years] — Full Analysis Set
  Years | 46.0 [18 to 83.0] | 46.0 [18.0 to 86.0] | 46.0 [18.0 to 86.0]
Age, Continuous [Mean (Standard Deviation); unit: Years] — Full Analysis Set
  Years | 46.3 (15.42) | 45.9 (14.99) | 46.1 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full Analysis Set
  Participants
    Female | 239 | 216 | 455
    Male | 213 | 235 | 448
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full Analysis Set
  Participants
    Hispanic or Latino | 230 | 238 | 468
    Not Hispanic or Latino | 222 | 213 | 435
    Not reported | 0 | 0 | 0
    Unknown | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full Analysis Set
  Participants
    American Indian or Alaska Native | 100 | 115 | 215
    Asian | 30 | 21 | 51
    Black or African American | 16 | 20 | 36
    Multiple | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Not reported | 21 | 21 | 42
    White | 285 | 274 | 559
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Full Analysis Set
  kg/m^2 | 28.9 (5.46) | 29.2 (6.56) | 29.0 (6.03)
Risk of Progression to Severe COVID-19 [Count of Participants; unit: Participants] — Risk of Progression to Severe COVID-19 is assessed based on participant's medical history - based on FDA/CDC guidelines. Summarized in the Full Analysis Set
  Participants
    High | 405 | 406 | 811
    Low | 47 | 45 | 92
Country [Count of Participants; unit: Participants]
  Argentina | 29 | 28 | 57
  Brazil | 7 | 12 | 19
  Czech Republic | 3 | 2 | 5
  Germany | 33 | 38 | 71
  Hungary | 2 | 1 | 3
  Italy | 37 | 33 | 70
  Japan | 26 | 14 | 40
  Mexico | 139 | 166 | 305
  Poland | 1 | 1 | 2
  Russian Federation | 55 | 51 | 106
  Spain | 31 | 37 | 68
  Ukraine | 5 | 10 | 15
  United Kingdom | 20 | 18 | 38
  United States | 64 | 40 | 104

OUTCOME MEASURES:

1. Primary Outcome: A Composite of Either Severe COVID-19 or Death From Any Cause Through Day 29
Description: Severe COVID-19 is characterized by a minimum of either pneumonia (fever, cough, tachypnea, or dyspnea, and lung infiltrates) or hypoxemia (SpO2 < 90% in room air and/or severe respiratory distress) and a WHO Clinical Progression Scale score of 5 or higher.
Time Frame: Baseline (Day 1) and Day 29
Population: Modified Full Analysis Set (mFAS) - All randomized participants who received IMP ≤ 7 days from symptom onset and were not hospitalized at baseline (≤ Day 1) for isolation purpose. For AZD7442, N = 413; Placebo, N = 421. For the analysis of the primary endpoint, only participants within this population who were assessed for the primary endpoint were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 410 | 419
Participants | 18 | 37
Statistical Analysis 1: Comparison: AZD7442 vs Placebo; AZD7442 vs Placebo; Test type: Superiority; p = 0.010, Cochran-Mantel-Haenszel; CMH was stratified by randomization factors; Relative Risk Reduction (100*[1-RR]) = 50.38, 95% CI 2-sided [14.38 to 71.25]

2. Secondary Outcome: A Composite of Death From Any Cause or Hospitalization for COVID-19 Complications or Sequelae Through Day 169
Description: Death from Any Cause or Hospitalization for COVID-19 Complications or Sequelae through Day 169
Time Frame: Baseline (Day 1) and Day 169
Population: Modified Full Analysis Set (mFAS) - All randomized participants who received IMP <= 7 days from symptom onset and were not hospitalized at baseline (<= Day 1) for isolation purpose. For AZD7442, N = 413; Placebo, N = 421. For the analysis of the Key Secondary Endpoint, only participants within this population who were assessed for the primary endpoint were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 404 | 411
Participants | 20 | 40
Statistical Analysis 1: Comparison: AZD7442 vs Placebo; AZD7442 vs Placebo; Test type: Superiority; p = 0.009, Cochran-Mantel-Haenszel; CMH was stratified by randomization factors; Relative Risk Reduction (100*[1-RR]) = 49.24, 95% CI 2-sided [14.72 to 69.79]

ADVERSE EVENTS:
Time Frame: From first dose of study drug until end of study, with an average of 436 days.
Description: AEs are reported for the Safety Analysis Set, defined as all participants randomized and dosed with IMP.
Arm/Group | AZD7442 | Placebo
All-Cause Mortality (participants affected / at risk) | 8/452 | 8/451
Serious Adverse Events (participants affected / at risk) | 46/452 | 65/451
Other Adverse Events (participants affected / at risk) | 230/452 | 224/451
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD7442 (N=452) | Placebo (N=451)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Superinfection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial diarrhoea (Infections and infestations) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 9 (9)
COVID-19 pneumonia (Infections and infestations) | 23 (23) | 37 (37)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Superior sagittal sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (2)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD7442 (N=452) | Placebo (N=451)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 8 (10) | 9 (9)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Decreased activity (General disorders) | 1 (1) | 0 (0)
Energy increased (General disorders) | 1 (1) | 2 (2)
Face oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 16 (16) | 15 (17)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 2 (2) | 2 (2)
Injection site haematoma (General disorders) | 1 (1) | 1 (1)
Injection site induration (General disorders) | 1 (1) | 0 (0)
Injection site inflammation (General disorders) | 1 (1) | 0 (0)
Injection site nodule (General disorders) | 1 (2) | 0 (0)
Injection site pain (General disorders) | 8 (12) | 11 (15)
Injection site swelling (General disorders) | 1 (2) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 1 (2)
Malaise (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 3 (4) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 3 (6) | 2 (3)
Vaccination site reaction (General disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (2) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Bed bug infestation (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 49 (49) | 43 (44)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 12 (12)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 2 (2)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (6) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Gonococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Gonorrhoea (Infections and infestations) | 0 (0) | 3 (3)
H3N2 influenza (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 4 (4) | 0 (0)
Influenza (Infections and infestations) | 4 (5) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 8 (10)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (2) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 2 (3)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 2 (2)
Post-acute COVID-19 syndrome (Infections and infestations) | 38 (39) | 29 (30)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 10 (11) | 9 (11)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral rhinitis (Infections and infestations) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 1 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 13 (29) | 13 (33)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 2 (2) | 0 (0)
Cardiac flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (2)
Nodal rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 2 (2)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Azygos lobe (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 3 (3)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 2 (2)
Diabetic retinal oedema (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (12) | 6 (6)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 4 (5)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 4 (4)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 1 (1)
Application site haematoma (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Injection site discomfort (General disorders) | 2 (3) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (2)
Genitourinary chlamydia infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 5 (7)
Syphilis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Hepatitis A antibody (Investigations) | 0 (0) | 1 (1)
Lipids abnormal (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 2 (2)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 7 (10) | 4 (5)
Dyslipidaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 9 (9) | 7 (7)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 8 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis enteropathic (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 10 (10)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mastication disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (5)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 2 (2) | 2 (2)
Amnesia (Nervous system disorders) | 2 (2) | 1 (1)
Anosmia (Nervous system disorders) | 8 (9) | 3 (3)
Apallic syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral hypoperfusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 8 (8) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 13 (14) | 11 (15)
Hemiparaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypergeusia (Nervous system disorders) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hyposmia (Nervous system disorders) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (2)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 4 (4)
Parosmia (Nervous system disorders) | 2 (2) | 3 (3)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Tarsal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (4)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bruxism (Psychiatric disorders) | 1 (1) | 0 (0)
Burnout syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (2)
Depression (Psychiatric disorders) | 5 (5) | 5 (5)
Insomnia (Psychiatric disorders) | 7 (7) | 2 (2)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 2 (2) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Bartholin's cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Breast discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial thickening (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 4 (4)
Hypomenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Polycystic ovaries (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 11 (12)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (8)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Unhealthy diet (Social circumstances) | 1 (1) | 0 (0)
Abdominal wall operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Brachiocephalic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 16 (16) | 18 (18)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Conjunctival disorder (Eye disorders) | 0 (0) | 1 (1)
Lymphostasis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of any part or entirely of study results requires prior written approval from sponsor, with no timeframe for sponsor to review.

DOCUMENTS (2):
  • Study Protocol (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT04723394/Prot_006.pdf
  • Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT04723394/SAP_007.pdf